CLINICAL TRIAL: NCT03485612
Title: Analysis of Change of Optic Nerve Sheath Diameter in in Patients Operated for Urological Reasons
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Tomasz Skladzien, senior assistant, Jagiellonian University
Other Study IDs: 1072.6120.30.2018
Record Dates: First submitted 2018-03-10; First posted 2018-04-02 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Anaesthetic Complication Neurological; Central Nervous System Depression
Keywords: Optic Nerve Sheath Diameter; Urological Anaesthesia; point of care USG

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- change of the optic nerve sheath diameter: The test group will be male and female patients, aged over 18 and below 90 years of age. Each patient will be operated for urological reasons in the position for lithotomy.
  Interventions: Diagnostic Test: Change of Optic Nerve Sheath Diameter

INTERVENTIONS:
Diagnostic Test: Change of Optic Nerve Sheath Diameter — In patients, the optic nerve sheath width (ONSD) examination will be performed twice: for the first time immediately after general anesthesia and again after surgery after placing the patient in a position on the back.

SUMMARY:
The assessment of the diameter of the optic nerve sheath (ONSD) using ultrasound can be a very helpful tool in the assessment of increased intracranial pressure in patients operated for urological procedures.

DETAILED DESCRIPTION:
Advantages of using ultrasound in the assessment of intracranial pressure:

simple, bedside examination, repetitive, generally available, cheap, no exposure to X-rays, no need to transport the patient to the CT laboratory

Differential diagnosis:

Widening of the size of the optic nerve sheath outside of increased intracranial pressure may occur in the following pathologies:

optic neuritis optic nerve injuries meningioma of the optic nerve arachnoid cyst around the optic nerve tumors of the cavernous sinus Blood edema may occur due to impaired blood flow. The research is to determine whether the patient's position for urological procedures is safe for the patients and whether as a result of staying in such a position there is no development of cerebral edema.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing urologic operation
* Adults 18 to 90 years of age
* American Society of Anesthesiologists Physical grade 1-3

Exclusion Criteria:

* Patients who did not agree to participate in the study
* Patients with ophthalmic diseases
* Patients with previous history of ophthalmic surgery
* Patients with neurological disorders
* Patients with history of head surgery due to neurological disorders
* Patients with history of disease with increased intracranial pressure
* Patients with history of disease with increased intraocular pressure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing urologic operation Adults 18 to 90 years of age American Society of Anesthesiologists Physical grade 1-3
Sampling Method: Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Optic Nerve Sheath Diameter | 10 hours

SECONDARY OUTCOMES:
neurological complications | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital in Cracow, Krakow, Poland

IPD SHARING:
Plan to Share IPD: No
We are undecided on this point.